CLINICAL TRIAL: NCT05757362
Title: Development of a Compliance Questionnaire for Therapeutic Home Exercise Program in Physiotherapy and Rehabilitation (CQ-HEPT) Using the Delphi Method
Brief Title: Development of Compliance Questionnaire for Home Exercise Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, Elif Elcin Dereli, Associate Proffessor, Istanbul Bilgi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 202240034145
Record Dates: First submitted 2022-12-26; First posted 2023-03-07 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Development, Consensus
Keywords: Delphi method; compliance; home exercise; questionnaire; validity; reliability
MeSH Terms: conditions — Patient Compliance | interventions — Physical Therapy Modalities; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Compliance Questionnaire for Therapeutic Home Exercise Program in Physiotherapy and Rehabilitation (Other): Participants will be asked to complete the questionnaire developed.
  Interventions: Other: Compliance Questionnaire for Therapeutic Home Exercise Program in Physiotherapy and Rehabilitation (cq-HEPT)

INTERVENTIONS:
Other: Compliance Questionnaire for Therapeutic Home Exercise Program in Physiotherapy and Rehabilitation (cq-HEPT) — An online application of the developed questionnaire form

SUMMARY:
Exercise is a valuable basic treatment method in the field of physiotherapy and rehabilitation. However, the effectiveness of exercise therapy requires the individual to be attentive, compliant, and disciplined. Therefore, it is important to examine the factors that may affect compliance with exercise. The main aim of this study is to develop a questionnaire that can describe individuals' compliance with participation in a home exercise program using the Delphi method and then analyze the psychometric validity and reliability of this questionnaire. The value that the evaluation questionnaire planned to be obtained at the end of such a study will add to exercise science, which is one of the most powerful treatment elements of physiotherapy and rehabilitation discipline, is important.

DETAILED DESCRIPTION:
Exercise is a valuable basic treatment method in the discipline of physiotherapy and rehabilitation. The importance of exercise in maintaining and improving health or in combating diseases and/or injuries has been recognized. However, exercise therapy requires care, compliance, and discipline, otherwise, it is not possible to achieve positive results from this type of treatment. Examining factors that affect adherence to exercise can help understand and resolve issues that may hinder individual participation. The planned aim of this study was to develop a questionnaire that could describe individuals' compliance with participation in a home exercise program using the Delphi method, and then analyze the psychometric validity and reliability of this questionnaire. For this reason, academic physiotherapists or physiotherapists with at least 5 years of clinical experience will be asked to identify questions and details that can assess individuals' compliance with home exercise. Based on their responses, a questionnaire with at least 10 questions will be prepared by the investigators. Then, the appropriateness of the questions of this questionnaire will be examined and presented to the expert opinions again. The participating experts will be asked to rate each item sent to them on a Likert-type scale of 1 (strongly disagree) to 5 (strongly agree) whether it should be included in the questionnaire. If there is 80% or more consensus on an item for 4 and 5, the item will be considered to have reached consensus. Once the questionnaire has been created based on the Delphi method, it will be administered as an online questionnaire to 50 volunteer participants who have been given a home exercise program within physiotherapy and rehabilitation treatment and thus the basic psychometric properties of the questionnaire (internal consistency, test-retest reliability) will be analyzed. The evaluation questionnaire planned to be obtained at the end of this study is expected to significantly contribute to the field of exercise science.

ELIGIBILITY:
Inclusion criteria for the Delphi rounds are individuals who meet at least one of the following criteria:

* Five or more years of professional experience in the field of Physiotherapy and Rehabilitation.
* Holding an academic position in the field of Physiotherapy and Rehabilitation.

For testing the obtained questionnaire,

The inclusion criteria are:

* To have recently or previously taken a home exercise program
* To be over 18 years old

The exclusion criteria are:

-To have a condition that prevents the individual from understanding and completing the online questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Compliance Questionnaire for Therapeutic Home Exercise Program in Physiotherapy and Rehabilitation (CQ-HEPT) | through study completion, an average of 6 months.
  The questionnaire planned to be developed by the investigators using the Delphi method

CONTACTS AND LOCATIONS:
Overall Officials: Elif E Dereli, Assoc. Prof., Study Chair — Istanbul Bilgi University; Tugba K Colak, Assoc. Prof., Study Director — Marmara University; Aycan C Reyhan, PhD, Principal Investigator — Istanbul Bilgi University; Cigdem Emirza, MSc, Principal Investigator — Istanbul Bilgi University
Locations (1):
- Istanbul Bilgi University, Istanbul, Beyoglu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Boynton PM, Greenhalgh T. Selecting, designing, and developing your questionnaire. BMJ. 2004 May 29;328(7451):1312-5. doi: 10.1136/bmj.328.7451.1312. PMID 15166072
- [Background] Jack B, Clarke AM. The purpose and use of questionnaires in research. Prof Nurse. 1998 Dec;14(3):176-9. PMID 10095687
- [Background] Lee J, Lee SH, Chang GT. Expert consensus on the development of a health-related questionnaire for the pediatric field of Korean medicine: a Delphi study. BMC Complement Med Ther. 2020 Jan 15;20(1):10. doi: 10.1186/s12906-019-2796-x. PMID 32020878
- [Background] Gagnon AJ, DeBruyn R, Essen B, Gissler M, Heaman M, Jeambey Z, Korfker D, McCourt C, Roth C, Zeitlin J, Small R; ROAM Collaboration. Development of the Migrant Friendly Maternity Care Questionnaire (MFMCQ) for migrants to Western societies: an international Delphi consensus process. BMC Pregnancy Childbirth. 2014 Jun 10;14:200. doi: 10.1186/1471-2393-14-200. PMID 24916892
- [Background] Antcliff D, Keeley P, Campbell M, Oldham J, Woby S. The development of an activity pacing questionnaire for chronic pain and/or fatigue: a Delphi technique. Physiotherapy. 2013 Sep;99(3):241-6. doi: 10.1016/j.physio.2012.12.003. Epub 2013 Feb 8. PMID 23395263
- [Background] Galloza J, Castillo B, Micheo W. Benefits of Exercise in the Older Population. Phys Med Rehabil Clin N Am. 2017 Nov;28(4):659-669. doi: 10.1016/j.pmr.2017.06.001. PMID 29031333
- [Background] Hotting K, Roder B. Beneficial effects of physical exercise on neuroplasticity and cognition. Neurosci Biobehav Rev. 2013 Nov;37(9 Pt B):2243-57. doi: 10.1016/j.neubiorev.2013.04.005. Epub 2013 Apr 25. PMID 23623982
- [Background] Gimenez-Meseguer J, Tortosa-Martinez J, Cortell-Tormo JM. The Benefits of Physical Exercise on Mental Disorders and Quality of Life in Substance Use Disorders Patients. Systematic Review and Meta-Analysis. Int J Environ Res Public Health. 2020 May 23;17(10):3680. doi: 10.3390/ijerph17103680. PMID 32456164
- [Background] de Labra C, Guimaraes-Pinheiro C, Maseda A, Lorenzo T, Millan-Calenti JC. Effects of physical exercise interventions in frail older adults: a systematic review of randomized controlled trials. BMC Geriatr. 2015 Dec 2;15:154. doi: 10.1186/s12877-015-0155-4. PMID 26626157
- [Background] Amatriain-Fernandez S, Murillo-Rodriguez ES, Gronwald T, Machado S, Budde H. Benefits of physical activity and physical exercise in the time of pandemic. Psychol Trauma. 2020 Aug;12(S1):S264-S266. doi: 10.1037/tra0000643. Epub 2020 Jun 1. PMID 32478537
- [Background] Moreno Reyes P, Munoz Gutierrez C, Pizarro Mena R, Jimenez Torres S. [Effects of physical exercise on sleep quality, insomnia, and daytime sleepiness in the elderly. A literature review]. Rev Esp Geriatr Gerontol. 2020 Jan-Feb;55(1):42-49. doi: 10.1016/j.regg.2019.07.003. Epub 2019 Oct 12. Spanish. PMID 31610889
- [Background] Nicolson PJA, Hinman RS, Wrigley TV, Stratford PW, Bennell KL. Self-reported Home Exercise Adherence: A Validity and Reliability Study Using Concealed Accelerometers. J Orthop Sports Phys Ther. 2018 Dec;48(12):943-950. doi: 10.2519/jospt.2018.8275. Epub 2018 Jul 27. PMID 30053792
- [Background] Newman-Beinart NA, Norton S, Dowling D, Gavriloff D, Vari C, Weinman JA, Godfrey EL. The development and initial psychometric evaluation of a measure assessing adherence to prescribed exercise: the Exercise Adherence Rating Scale (EARS). Physiotherapy. 2017 Jun;103(2):180-185. doi: 10.1016/j.physio.2016.11.001. Epub 2016 Nov 9. PMID 27913064
- [Background] A brief history of RAND [Internet]. Rand.org. [cited 2022 Dec 26]. Available from: https://www.rand.org/about/history.html
- [Background] Dalkey N, Helmer O. An experimental application of the DELPHI method to the use of experts. Manage Sci [Internet]. 1963;9(3):458-67. Available from: http://dx.doi.org/10.1287/mnsc.9.3.458